CLINICAL TRIAL: NCT04604899
Title: A Phase 2 Study of the Safety of Repeat Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects With Retinitis Pigmentosa (RP)
Brief Title: Safety of Repeat Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects With Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: jCyte, Inc (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JC02-2
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Retreated subjects (Experimental): Subjects receiving human retinal progenitor cells (jCell) who have previously received jCell is a jCyte study.
  Interventions: Biological: human retinal progenitor cells

INTERVENTIONS:
Biological: human retinal progenitor cells — single intravitreal injection of 6.0 million human retinal progenitor cells (hRPC)
  Other Names: jCell

SUMMARY:
The primary objective of the study is to assess the safety of repeat injection of human retinal progenitor cells (jCell) in adult subjects with RP that have previously been treated with jCell.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, Phase 2 study of human retinal progenitor cells (jCell) for the treatment of retinitis pigmentosa (RP). The study will include only subjects previously treated with jCell.

To assess reinjection of a previously treated eye, subjects who have previously been treated with jCell and desire a second treatment in the same eye will be enrolled. Subjects must have completed at least 12 months of follow up since the prior injection of jCell. Subjects who have had both eyes previously treated with jCell will only have one eye retreated; the eye to be retreated will preferably be the better seeing eye, but exceptions may be made by the study investigator, taking into consideration BCVA, prior response to treatment, and any other medical conditions that may indicate which eye is the best candidate for retreatment. Subjects will be followed for 12 months for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give written informed consent, able to make the required study visits and follow study protocol instructions.
2. Completed the 12 months of follow up in the subject's most recent jCell study and did not withdraw from the study for any reason.
3. Adequate organ function:

   * blood counts (hematocrit, Hgb, WBC, platelets and differential) within normal range, or if outside of normal range, not clinically significant as judged by the investigator
   * liver function: alanine transaminase [ALT] and aspartate transaminase [AST] ≤2 times the upper limit of the normal range
   * total bilirubin ≤1.5 times the upper limit of the normal range
   * renal function: serum creatinine ≤1.25 times the upper limit of the normal range
4. A female patient of childbearing potential (not surgically sterilized and less than one year postmenopausal) must have a negative pregnancy test (urine human chorionic gonadotropin) at entry (prior to injection) and must have used medically accepted contraception for at least one month prior to treatment. Women of childbearing potential and men must be advised to use a medically accepted method of contraception for at least 12 months following treatment.

Exclusion Criteria:

1. Malignancy, end-stage major organ disease (heart failure, significant arrhythmias, stroke or transient ischemic attacks, diabetes, immunosuppressive or autoimmune state, major psychiatric disorder, epilepsy, thyroid disease, COPD, renal failure, or any chronic systemic disease requiring continuous treatment with systemic steroids, anticoagulants or immunosuppressive agents.
2. History of eye disease other than RP that impairs visual function, including retinal vascular disease, elevated intraocular pressure/glaucoma, severe posterior uveitis, clinically significant macular edema, media opacity precluding visual exam, amblyopia and/or longstanding constant strabismus, as well as patients who require other intravitreal therapies
3. Allergy to penicillin or streptomycin.
4. Adverse reaction to DMSO.
5. Unable or unwilling to undergo pupil dilation, topical anesthesia or any protocol-required procedure.
6. Women who are nursing or who are planning to nurse during the 12 months that would follow study treatment.
7. Any circumstance that in the opinion of the investigator, would interfere with participation in, or compliance with the study protocol
8. Treatment with corticosteroids (systemic, periocular or intravitreal) or any other non-approved, experimental, investigational or neuroprotectant therapy (systemic, topical, intravitreal) in either eye within 90 days of planned second injection.
9. Cataract surgery within three months prior to treatment or anticipated to need cataract surgery within a year of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitul Mehta, MD, Principal Investigator — University of California, Irvine/Gavin Herbert Eye Institute; David Liao, MD, Principal Investigator — Retina-Vitreous Associates Medical Group, Los Angeles CA; Anthony Jospeh, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (3):
- United States (3):
  - Gavin Herbert Eye Inst, Univ Cal Irvine, Irvine, California
  - Retina-Vitreous Associates Medical Group, Los Angeles, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retreated Subjects
Started | 30
Completed | 23
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 170.14 (9.856)
Weight [Mean (Standard Deviation); unit: kg] | 84.00 (24.387)
Study eye [Count of Participants; unit: Participants]
  Right (OD) | 14
  Left (OS) | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intravitreal Injection of hRPC
Description: Assessed by percentage of subjects with treatment emergent adverse events
Time Frame: 12 months
Population: Safety population: all subjects who receive any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 30
Participants
  Subjects with any TEAEs | 15
  Subjects with any TEAEs related/possibly related to study drug | 6
  Subjects with any serious TEAEs | 6
  Subjects with any serious TEAEs related/possibly related to study drug | 2
  Subjects with any severe TEAEs related/possibly related to study drug | 1

2. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Mean change in BCVA in study eye from baseline to month 12 as assessed by E-ETDRS. A letter score is used to compare change over time, with a higher number of letters representing better visual function, and a lower number of letters representing worse visual function. For example, 85 letters is equivalent to 20/20 visual acuity and 5 letters is equivalent to 20/800 visual acuity. A change value is derived for each subject by taking the letter score at 12 months and subtracting the letter score at baseline. A mean of all change values is then calculated.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: letters correct
Groups:
- Retreated Subjects: Subjects receiving human retinal progenitor cells (jCell) who have previously received jCell in a jCyte study.
  human retinal progenitor cells: single intravitreal injection of 6.0 million human retinal progenitor cells (hRPC)
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 23
letters correct | -2.340 (5.8963)

3. Secondary Outcome: Kinetic Visual Field Area
Description: Mean change in total kinetic visual field (KVF) area (degrees squared) of all islands of vision from baseline to 12 months. The Octopus 900 will be used for KVF testing using a specified target of V4e for subjects with a more severely impaired visual field (<10,000deg2) and a target of III4e and I4e for better seeing subjects (>10,000deg2). Target size is selected based on the Baseline visit. Whatever target size(s) is/are selected, the same size will be used throughout the study on that particular eye for that particular patient.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: degrees squared
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 23
degrees squared | -493.96 (1268.067)

4. Secondary Outcome: Contrast Sensitivity (Peak)
Description: Contrast sensitivity (CS) measures the ability of a subject to distinguish between finer and finer increments of light versus dark (contrast), as measured with a vertical striped pattern that varies in stripe width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each size of the target (i.e., at various CPDs). A CS curve is created by using the threshold of CS means at each target size, with the highest or most sensitive value (regardless of the CPD) representing the peak of the curve (i.e., peak contrast sensitivity). The unit of measure is therefore the peak contrast sensitivity regardless of the target size (i.e., CPD) being used to perform the measurement. The higher the value, the better the ability to detect contrast. The data shown here represent the mean change from Baseline to 12 months in the subjects' peak of the CS curve.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Arbitrary Units (AU)
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 16
Arbitrary Units (AU) | -0.57 (6.690)

5. Secondary Outcome: Low Luminance Mobility Test (LLMT)
Description: The LLMT identifies the performance of patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to a bright indoor room (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest light level of 0 lux (completely dark room) corresponds to a scale score of 13, whereas the brightest light level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement in low light vision, whereas a negative scale score change represents a decline in low light vision.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Retreated Subjects
Number analyzed (Participants) | 21
scores on a scale | -0.1 (1.96)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Retreated Subjects (All Ocular AEs Were Reported in Study Eyes): Subjects receiving human retinal progenitor cells (jCell) who have previously received jCell is a jCyte study.
  human retinal progenitor cells: single intravitreal injection of 6.0 million human retinal progenitor cells (hRPC)
Arm/Group | Retreated Subjects (All Ocular AEs Were Reported in Study Eyes)
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retreated Subjects (All Ocular AEs Were Reported in Study Eyes) (N=30)
Tractional retinal detachment (Eye disorders) | 1 (1)
Vitreoretinal traction syndrome (Eye disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Hallucination (Psychiatric disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retreated Subjects (All Ocular AEs Were Reported in Study Eyes) (N=30)
Conjunctival haemorrhage (Eye disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04604899/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04604899/SAP_001.pdf